CLINICAL TRIAL: NCT00908401
Title: Breastmilk or Oral Sucrose Solution in Preterm Neonates for Procedural Pain: a Randomized, Controlled Study
Brief Title: Analgesic Effect of Breastmilk for Procedural Pain in Preterm Infants
Acronym: BMoS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Centre Hospitalier Intercommunal de Creteil, Centre Hospitalier Intercommunal de Creteil
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHICreteil
Record Dates: First submitted 2009-05-22; First posted 2009-05-25 (Estimated); Last update posted 2009-05-25 (Estimated); Status verified 2009-05

CONDITIONS: Procedural Pain
Keywords: breastmilk; oral sucrose; analgesia; preterm neonates; Neonates
MeSH Terms: conditions — Pain, Procedural; Agnosia | interventions — Sucrose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- sucrose (Active Comparator): This group will receive oral sucrose for procedural pain
  Interventions: Other: Oral Sucrose
- breastmilk (Experimental): this group will receive breastmilk as analgesic product to avoid procedural pain
  Interventions: Other: Breastmilk

INTERVENTIONS:
Other: Breastmilk — Breastmilk: 0.2 ml
  Arms: breastmilk
Other: Oral Sucrose — oral sucrose: 0.2 ml one time 1 minute before the painful procedure with a pacifier
  Arms: sucrose

SUMMARY:
Hypothesis: Breastmilk has a more powerful analgesic effect than oral sucrose to avoid procedural pain in preterm neonates.

The objective is to test this hypothesis in a randomized, controlled study using a standardized and validated pain scale (DAN). The sample size is 21 preterm infants in each two groups. The main end point is a reduction of the risk to have a DAN superior to 1 from 80% with oral sucrose to 40% with breastmilk.

ELIGIBILITY:
Inclusion Criteria:

* preterm neonates born before 27 and 29+6 weeks GA
* blood sampling procedure
* obtention of parental consent

Exclusion Criteria:

* congenital malformation
* intravenous continuous analgesia
* contraindications to feed
* high grade intracerebral hemorrhage

Ages: 3 Days to 10 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Estimated)
Dates: Start 2009-04; Primary Completion 2009-07 (Estimated); Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
Decrement from 80 to 40% of frequency of DAN's scale score superior to 1 using breastmilk instead of oral sucrose | One time during day 3 or 4 then day 7 to 10

CONTACTS AND LOCATIONS:
Overall Officials: Elodie Zana, MD, Principal Investigator — Centre Hospitalier Intercommunal Creteil
Locations (1):
- Centre Hospitalier Intercommunal de Creteil, Créteil, France

REFERENCES:
- [Background] Schollin J. Analgesic effect of expressed breast milk in procedural pain in neonates. Acta Paediatr. 2004 Apr;93(4):453-5. doi: 10.1080/08035250410027959. PMID 15188969
- [Background] Carbajal R, Veerapen S, Couderc S, Jugie M, Ville Y. Analgesic effect of breast feeding in term neonates: randomised controlled trial. BMJ. 2003 Jan 4;326(7379):13. doi: 10.1136/bmj.326.7379.13. PMID 12511452
- [Background] Carbajal R, Paupe A, Hoenn E, Lenclen R, Olivier-Martin M. [APN: evaluation behavioral scale of acute pain in newborn infants]. Arch Pediatr. 1997 Jul;4(7):623-8. doi: 10.1016/s0929-693x(97)83360-x. French. PMID 9295899